CLINICAL TRIAL: NCT06169592
Title: Verification of Prognostic Risk Factors of Thrombohemorrhagic Complications in Early Follow-up Period in Recipients After Living Related Liver Transplantation
Brief Title: Verification of Risk Factors of Thrombohemorrhagic Complications in Recipients After Related Liver Transplantation
Acronym: VORTAL
Status: Recruiting | Type: Observational
Sponsor: Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov (Other)
Responsible Party: Principal Investigator, Azam Babadjanov, Professor, Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov
Other Study IDs: 05122023
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-07

CONDITIONS: Liver Cirrhosis; Liver Transplant; Complications
MeSH Terms: conditions — Liver Cirrhosis | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver transplant group
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Related transplantation of the right lobe of the liver

SUMMARY:
The aim of the study is to improve the results of related transplantation of the right liver lobe by verifying the general predictors of the development of hemostatic system disorders and optimizing a comprehensive program for thrombohemorrhagic complications preventing.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and up to 70 years;
* Signed informed consent for inclusion to the study;
* End stage liver cirrhosis.

Exclusion Criteria:

* Pregnancy;
* Extrahepatic factors influencing systemic hemostasis;
* Concomitant hematological diseases affecting the hemostatic system;
* Severe concomitant disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage liver cirrhosis who underwent living related liver transplantation.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Thrombosis of vascular anastomosis | 1 month
  Thrombosis of arterial or venous anastomosis after intervention

SECONDARY OUTCOMES:
Hemorrhagic complications | 1 month
  Any hemorrhagic complications after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Republican specialized scientific and practical medical center of surgery named after academician V.Vakhidov, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided